CLINICAL TRIAL: NCT05948722
Title: Behavioral Intervention Program Based on Motivational Interview to Improve Oral Hygiene in Adults - a Randomized Clinical Trial
Brief Title: Behavioral Intervention Program Based on Motivational Interview
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Carlos Heitor Cunha Moreira, Principal Investigator, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 059082
Record Dates: First submitted 2023-05-02; First posted 2023-07-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Periodontal Diseases; Motivational Interviewing
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Interview Group (MIG) (Experimental): Participants assigned to this arm will complete three to five MI sessions
  Interventions: Behavioral: Motivational Interview Group (MIG)
- Conventional treatment group (CTG) (Active Comparator): Participants assigned to this arm will receive the conventional treatment
  Interventions: Procedure: Conventional treatment group (CTG)

INTERVENTIONS:
Behavioral: Motivational Interview Group (MIG) — Brief MI intervention with the conventional treatment
  Arms: Motivational Interview Group (MIG)
Procedure: Conventional treatment group (CTG) — Conventional treatment
  Arms: Conventional treatment group (CTG)

SUMMARY:
The best way for dental professionals act using dialogue methods and individual approaches in daily clinical practice to change behavioral is still inconclusive. Thus, the objective will be evaluate the effect of using motivational interviewing as part of the treatment of periodontitis in order to increase the adherence of adults to adequate oral health behavior.

DETAILED DESCRIPTION:
Patient-related approaches may show better results in treatment of periodontal diseases. The best way for the dental surgeon to act using these methods is still inconclusive. The aim of this study is to evaluate the effectiveness of using motivational interviewing as part of the treatment of periodontitis in order to increase adult adherence to adequate oral health behavior. A randomized clinical trial, with a sample size of at least 72 subjects, >18 years of age and with at least 18 teeth, will be investigated. Individuals in the test group will receive a collaborative communicative approach, inspired by the motivational interview, while the control group will receive the information/instructions in a conventional approach. The efficacy variables for evaluating the pattern of self-control of periodontal infection will be the bleeding on probing (BoP), gingival index (GI, primary efficacy variable), the plaque index (PI) and patient-based outcomes will be assessed using quality of life questionnaires. Additionally, questionnaires will be applied to obtain sociodemographic, behavioral and self-perception of oral health data. Univariate and multivariate analyzes will be performed and conducted in the Statistical Products Service Solutions software (SPSS, version 25). Thus, it will be possible to assess whether brief oral health education interventions centered on the individual can be used by dental surgeons in order to effectively improve oral hygiene behaviors in adults, obtaining better clinical results and a better quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults, over 18-year-old;
* BoP (Bleeding on probing) in at least 30% of sites;
* Diagnosed periodontitis.

Exclusion Criteria:

* Smoking;
* Diabetes;
* Pregnancy (or the planning of pregnancy);
* Immunosuppressive illness or a medication, hepatitis, HIV, a bleeding illness or a anticoagulant;
* A need for the antibiotic prophylaxis;
* Hyposalivation or use of medications that cause hyposalivation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in Bleeding on Probing to evaluate the improvement in hygiene behavior | baseline, 15 days after supragingival treatment, 30 and 60 days after subgingival treatment and through study completion, an average of 1 year
  BoP - Dichotomic response after probing the gingival sulcus. High values mean worst condition.
The change in Plaque Index to evaluate the improvement in hygiene behavior | baseline, 15 days after supragingival treatment, 30 and 60 days after subgingival treatment and through study completion, an average of 1 year
  PI - Each of the 6 sites of the tooth is given a score from 0 to 3. High values mean worst condition.
The change in Gingival index to evaluate the improvement in hygiene behavior | baseline, 15 days after supragingival treatment, 30 and 60 days after subgingival treatment and through study completion, an average of 1 year
  GI - Each of the 6 sites of the tooth is given a score from 0 to 3. High values mean worst condition.
Patient satisfaction assessed by the change in Quality of Life questionnaire | baseline, 60 days after subgingival treatment and through study completion, an average of 1 year
  Quality of life - % of patients with better scores (lowest values) of quality of life. It can vary from 0 to 56.
Patient perception assessed by the change in autoperception of oral health questionnaire | baseline, 60 days after subgingival treatment and through study completion, an average of 1 year
  Autoperception of oral health - rate of patients with better condition of oral health perception. The answer options are: Great; Good; Regular; Bad; Terrible. 0-4 (lower scores mean better self-perception).

SECONDARY OUTCOMES:
Oral hygiene-related self-efficacy assessed by the oral hygiene-related selfefficacy (OHSE) questionnaire | 60 days after subgingival treatment and six months later
  Oral hygiene-related self-efficacy: % of patients with higher scores of self-efficacy. It ranges from 19 to 76, higher scores mean better self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Heitor Moreira, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No